CLINICAL TRIAL: NCT07132853
Title: Assessment of Physical Activity Levels in Patients With Cardiac Arrhythmias
Acronym: PAL-PAC
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Savia Christina Pereira Bueno, Principal Investigator, University of Sao Paulo
Other Study IDs: 5.127.777
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Arrhythmia; Physical Activity
Keywords: arrythmia; physical activity
MeSH Terms: conditions — Arrhythmias, Cardiac; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arrhythmia: Physical activity level description

SUMMARY:
Physical activity is defined as any bodily movement that results in energy expenditure. Athletes are individuals who engage in planned, structured physical exercise under guidance, with specific goals and competitive objectives. For this population, pre-participation cardiovascular screening is well established, aiming to identify cardiac conditions that may lead to sudden death and/or cardiovascular events. However, athletes represent a minority of patients attending cardiac arrhythmia outpatient clinics. Most patients are either sedentary or engage in-or wish to engage in-some form of physical activity, but are often discouraged for various reasons, leading to increased physical inactivity. This occurs despite the well-documented benefits of physical activity across all age groups and various forms of heart disease, including improved quality of life, reduced depression and anxiety, and enhanced overall well-being. Despite existing recommendations, the prevalence of physically active individuals among patients followed at the Arrhythmia Outpatient Clinic of the Heart Institute (InCor) of the Hospital das Clínicas, University of São Paulo, remains unknown. Understanding these factors through such mapping may contribute to improved clinical management and potentially enhance the quality of life of patients with cardiac arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a documented diagnosis of arrhythmia who are followed at the arrhythmia outpatient clinic of InCor.
2. Signed informed consent form or assent form.

Exclusion Criteria:

1. Bedridden patients or those with mobility impairments.
2. Patients with advanced-stage diseases (estimated life expectancy of less than one year).
3. Patients participating in other studies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 100 consecutive patients followed at the arrhythmia outpatient clinic of InCor - HCFMUSP.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
SF-12 Health Survey | Baseline
  Quality of life was assessed using SF-12's Physical and Mental scores.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Baseline
  Describe the physical activity level by IPAQ

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil